CLINICAL TRIAL: NCT00807300
Title: Phase-III-Study to Evaluate the Efficacy of CT-guided Brachytherapy Versus Transarterial Chemoembolization in Patients With Unresectable Hepatocellular Carcinoma.
Brief Title: Computed Tomography (CT) - Guided Brachytherapy Versus Transarterial Chemoembolization in Patients With Unresectable Hepatocellular Carcinoma
Acronym: CEAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Jens Ricke, Prof. Jens Ricke, University of Magdeburg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005-000569-21
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: percutaneous treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- brachytherapy (Active Comparator)
  Interventions: Radiation: CT-guided brachytherapy
- TACE (Other): transarterial chemoembolization
  Interventions: Procedure: transarterial chemoembolization

INTERVENTIONS:
Radiation: CT-guided brachytherapy — catheter placed into the tumor by CT-guidance, radiation with iridium 192
  Arms: brachytherapy
Procedure: transarterial chemoembolization — application of doxorubicin and cisplatin in lipiodol into the tumor-feeding artery
  Arms: TACE

SUMMARY:
Percutaneous, image-guided tumor ablation has evolved as a genuine alternative for the treatment of unresectable hepatocellular carcinoma. Published data exploring stereotactic or proton beam percutaneous irradiation have revealed,that hepatocellular carcinoma (HCC) is radiosensitive to certain protocols. In Phase I and II studies, the investigators investigated the potential role of local irradiation in primary and secondary liver tumors employing a Iridium192 source. The promising results of previous studies indicate that CT-guided brachytherapy might play a role in the treatment of unresectable HCC.

Therefore, the investigators started a randomized, controlled, clinical Phase-II study to evaluate the efficacy and survival-benefits of brachytherapy versus transarterial chemoembolization in patients with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HCC by histopathology or according to the criteria of the Consensus Conference of the European Association for the Study of Liver Disease
* unresectable HCC
* Karnofsky-Index > 70
* estimated life expectancy > 16 weeks
* adequate bone marrow function
* adequate contraception for female patients
* informed consent

Exclusion Criteria:

* portal vein thrombosis on the tumor side
* extrahepatic spread
* Child C
* other untreated malignant disease
* general contraindication for chemotherapy
* active infectious disease
* neuropathy, platin-allergy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to untreatable progression | the follow up period

SECONDARY OUTCOMES:
Time to progression | the follow up period
Overall survival | the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ricke, M.D., Principal Investigator — Clinic of Diagnostic Radiology and Nuclear Medicine, University Magdeburg
Locations (1):
- Clinic of Diagnostic Radiology and Nuclear Medicine, Medical Faculty, University Magdeburg, Magdeburg, Saxony-Anhalt, Germany